CLINICAL TRIAL: NCT02048982
Title: What Influences Physicians' Decisions - Statistics or Stories?
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Bishop_stats_stories
Record Dates: First submitted 2014-01-27; First posted 2014-01-29 (Estimated); Last update posted 2018-09-12 (Actual); Status verified 2018-09

CONDITIONS: Prescribing Tendencies
Keywords: physician prescribing; behavioral economics; primary care practice
MeSH Terms: interventions — Guidelines as Topic; Costs and Cost Analysis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Guideline and Cost (Experimental): The Choosing Wisely guideline and the cost of the test at our institution: $60.35 for a basic metabolic panel.
  Interventions: Behavioral: Guideline; Behavioral: Cost
- Guideline (Placebo Comparator): The Choosing Wisely guideline: "Don't perform blood chemistry panels in asymptomatic, healthy adults."
  Interventions: Behavioral: Guideline
- Guideline and Victim (Active Comparator): The Choosing Wisely Guideline and a clinical scenario with a patient as an identifiable victim who suffered harm from having an unnecessary test done
  Interventions: Behavioral: Guideline; Behavioral: Victim
- Guideline, Cost, and Victim (Experimental): The Choosing Wisely guideline and a clinical scenario with a physician as an identifiable victim who suffered harm when he ordered an unnecessary test.
  Interventions: Behavioral: Guideline; Behavioral: Cost; Behavioral: Victim

INTERVENTIONS:
Behavioral: Guideline — Physicians will receive information on the Choosing Wisely Guideline
Behavioral: Cost — Physicians will receive cost information.
  Arms: Guideline and Cost; Guideline, Cost, and Victim
Behavioral: Victim — Physicians will receive information on an identifiable victim.
  Arms: Guideline and Victim; Guideline, Cost, and Victim

SUMMARY:
The purpose of this study is to test whether physicians change their use of non-recommended tests, procedures, or medications more in response to evidence based-guidelines, price information, or an individual patient's story.

DETAILED DESCRIPTION:
We will perform a randomized controlled trial (RCT) of information presented to physicians to test the hypothesis that an identifiable victim affects physician practice behavior more than a statistical victim.

Specifically, we will answer the following research questions: 1) do physicians order fewer non-recommended tests, procedures, or medications if they are told about a patient or a physician who had a bad outcome from that test, procedure, or medication than if they are simply told the guideline or the cost of the test, procedure or medication, 2) does the effect of learning about the identifiable victim last longer than the effect of learning about the guideline or the cost of a test, procedure, or medication, and 3) does the identifiable victim effect differ if the victim is a patient or a physician? We hypothesize that because of the propensity to respond more to the identifiable victim rather than the statistical victim that physicians will order fewer unnecessary tests when they are told about an individual patient case than if they are simply told about the guideline, that the effect of the identifiable victim will last longer than the effect of the statistical victim, and that a patient as the identifiable victim will have more effect than a physician as the identifiable victim.

The identifiable victim effect refers to the tendency to offer more aid to a specific, identifiable victim rather than a vaguely defined group of people with the same need. In the this study, the identifiable victim is a fictional patient who experience a negative consequence as a result of an unnecessary test. The identifiable victim effect is described and studied in the following articles:

Small D. Sympathy and callousness: The impact of deliberative thought on donations to identifiable and statistical victims. Organizational Behavior and Human Decision Processes 2007;102:143-53.

George Loewenstein, Deborah A. Small, and Jeff Strand. "Statistical, identifiable, and iconic victims" in Edward J. McCaffery, Joel Slemrod (2006). Behavioral public finance. Russell Sage Foundation; pp. 32-35.

ELIGIBILITY:
Inclusion Criteria:

* Primary care physicians in the Weill Cornell Physicians Organization

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Percentage of blood chemistry tests among visits by adult patients under 65 | Within 1 week of receiving the intervention
Percentage of blood chemistry tests among visits by adult patients under 65 | Within 1 month of receiving the scenario

SECONDARY OUTCOMES:
Physicians' attitudes and perceived practice immediately after reading the scenario | Immediate (up to 5 min)

CONTACTS AND LOCATIONS:
Locations (1):
- Weill Cornell Medical College, New York, New York, United States